CLINICAL TRIAL: NCT02317913
Title: Epidemiologic Features of Kawasaki Disease in Shanghai From 2008 Through 2012
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Fudan University (Other)
Collaborators: Shanghai Children's Medical Center (Other); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); Ruijin Hospital (Other); Shanghai 6th People's Hospital (Other); Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other); Changhai Hospital (Other); Shanghai Tongji Hospital, Tongji University School of Medicine (Other)
Responsible Party: Principal Investigator, Guoying huang, Professor,President, Children's Hospital of Fudan University
Other Study IDs: kd2008-2012
Record Dates: First submitted 2014-12-08; First posted 2014-12-17 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2015-03

CONDITIONS: Kawasaki Disease
Keywords: Kawasaki disease; Epidemiology; Incidence; Coronary arterial lesions; Shanghai
MeSH Terms: conditions — Mucocutaneous Lymph Node Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
To investigate the epidemiological pictures of Kawasaki disease (KD) in Shanghai from 2008 through 2012, and illustrate the risk factors of coronary arterial lesions .

DETAILED DESCRIPTION:
A questionnaire form and diagnostic guidelines for KD will be sent to 50 hospitals providing pediatric medical care in Shanghai, China. All patients with KD diagnosed during January 2008 through December 2012 will be recruited and analyzed. Distribution of age at onset and seasonal features of disease incidence wil be described. Univariate and multivariate association analyses will be performed to identify risk factors to Coronary arterial lesions (CAL) defined as ectasia or aneurysm by using multivariate logistic regression model.

ELIGIBILITY:
Inclusion Criteria:

* The 5th revised edition of diagnostic criteria for KD, issued by the Japan Kawasaki Disease Research Committee at the 7th International Kawasaki Disease Symposium in 2002, was adopted. Cases were included in the study if the patients had at least five of the following six clinical manifestations or at least four signs together with coronary abnormalities documented by echocardiography or coronary angiography:

  1. fever persisting 5 days or longer (inclusive of those cases in whom the fever has subsided before the 5th day in response to therapy)
  2. bilateral conjunctival congestion
  3. changes of lips and oral cavity, such as reddening of lips, strawberry tongue, diffuse congestion of oral and pharyngeal mucosa
  4. polymorphous exanthema
  5. changes of peripheral extremities, such as reddening of palms and soles, indurative edema at initial stage, or membranous desquamation from fingertips at convalescent stage
  6. acute nonpurulent cervical lymphadenopathy. In addition, the cases of incomplete KD, diagnosed with referring to the guidelines for incomplete KD made by American Academy of Pediatrics (AAP) and American Heart Association (AHA) in 2004, were also included in this investigation

     Exclusion Criteria:
* The cases were not in accordance with the recruited criteria

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: All patients with KD diagnosed during January 2008 through December 2012 in Shanghai
Sampling Method: Non-Probability Sample
Enrollment: 2402 (Actual)
Dates: Start 2013-04; Primary Completion 2015-11 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
incidence of coronary artery lesions(CAL) | 5 years
  according to the result of the echocardiography performed in the acute phase ,early and late recovery of Kawasaki disease

CONTACTS AND LOCATIONS:
Locations (1):
- Children Hospital of Fudan University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Chen JJ, Ma XJ, Liu F, Yan WL, Huang MR, Huang M, Huang GY; Shanghai Kawasaki Disease Research Group. Epidemiologic Features of Kawasaki Disease in Shanghai From 2008 Through 2012. Pediatr Infect Dis J. 2016 Jan;35(1):7-12. doi: 10.1097/INF.0000000000000914. PMID 26372452